CLINICAL TRIAL: NCT00644254
Title: The Prognostic Impact of Extracapsular Lymph Node Involvement (ECLNI) in Ductal Pancreatic Adenocarcinoma (DPAC).
Brief Title: The Prognostic Impact of Extracapsular Lymph Node Involvement in Ductal Pancreatic Adenocarcinoma
Acronym: ECLNI DPAC
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Other Study IDs: ECLNI DPAC
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Pancreatic Neoplasms; Pancreatic Adenocarcinoma
Keywords: Prognosis; Extracapsular lymph node involvement
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Resected DPAC: 145 consecutive resections for primary ductal pancreatic adenocarcinoma (DPAC)performed between 1998 and 2005.
  Interventions: Procedure: Pancreatic resection

INTERVENTIONS:
Procedure: Pancreatic resection — PPPD, Whipple, Total pancreatectomy or left pancreatectomy.

SUMMARY:
Extracapsular lymph node involvement (ECLNI) has been identified as a pathological variable associated with worse outcome in esophageal, gastric and colorectal cancer. No studies so far have studied its prognostic impact in ductal pancreatic adenocarcinoma (DPAC). The goal of the investigators is to determine the prognostic value of ECLNI in a prospective consecutive series of 145 patients with DPAC, who underwent resection of their primary tumor between 1998 and 2005.

DETAILED DESCRIPTION:
Presence and extent of extracapsular lymph node involvement (ECLNI) will be scored by reviewing all original pathological slides.

ECLNI is defined as metastatic adenocarcinoma extending through the nodal capsule into the perinodal fatty tissue.

Observers: 1 experienced board-certified GI pathologist, blinded for follow-up results.

Follow-up data are obtained by reviewing patients charts and by a telephone survey of the patient's GP/gastroenterologist in November 2007.

Statistical analysis:

* Common closing date: 1/11/2007
* Kaplan-Meier survival analysis (Log-Rank, Wilcoxon)
* Cox logistic regression (uni/multivariate)

ELIGIBILITY:
Inclusion Criteria:

* DPAC
* Primary resection

Exclusion Criteria:

* Positive section margins
* non DPAC, other tumor
* Postoperative mortality
* Neoadjuvant chemo/radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Resected ductal pancreatic adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Overall cancer-specific survival | 11/2007

SECONDARY OUTCOMES:
Disease-free survival (DFS)& Correlation of ECLNI with other pathological variables | 11/2007

CONTACTS AND LOCATIONS:
Overall Officials: Baki Topal, MD, PhD, Study Director — Catholic University Leuven (KULeuven), Belgium; Gregory Sergeant, MD, Principal Investigator — Catholic University Leuven, Belgium; Nadine Ectors, MD, PhD, Principal Investigator — Catholic University Leuven, Belgium
Locations (1):
- Department of Abdominal Surgery, Leuven, Vlaams-Brabant, Belgium